CLINICAL TRIAL: NCT01468961
Title: Pilot Study of Internet-based Cognitive Behavior Therapy for Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Brjann Ljotsson, Associate professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIBRO-P
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Internet-based CBT (Experimental)
  Interventions: Behavioral: Internet-based CBT

INTERVENTIONS:
Behavioral: Internet-based CBT — 10 weeks of internet-based CBT with online therapist contact

SUMMARY:
This pilot trial will include 30-40 participants with a diagnosis of fibromyalgia. The purpose of the study is to evaluate an internet-based treatment protocol based on cognitive behavioral therapeutic principles. Participants are required to have a previous diagnosis of fibromyalgia before entering into the trial. The treatment will be 10 weeks long and all included participants will be given treatment, i.e. there is no randomization to a comparison group.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of fibromyalgia

Exclusion Criteria:

* Current diagnosis of severe psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The Fibromyalgia Impact Questionnaire | Once, 1 week before start of treatment
The Fibromyalgia Impact Questionnaire | Once, immediately after treatment
The Fibromyalgia Impact Questionnaire | Once, 6 months after treatment

SECONDARY OUTCOMES:
Short form 12-item Questionnaire | Once, 1 week before start of treatment
Short form 12-item Questionnaire | Once, immediately after treatment
Short form 12-item Questionnaire | Once, 6 months after treatment
Hospital Anxiety and Depression Scale | Once, 1 week before start of treatment
Hospital Anxiety and Depression Scale | Once, immediately after treatment
Hospital Anxiety and Depression Scale | Once, 6 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Department of Clinical Neuroscience, Section of psychiatry, Karolinska Hospital Solna R5, Stockholm, Sweden

REFERENCES:
- [Result] Ljotsson B, Atterlof E, Lagerlof M, Andersson E, Jernelov S, Hedman E, Kemani M, Wicksell RK. Internet-delivered acceptance and values-based exposure treatment for fibromyalgia: a pilot study. Cogn Behav Ther. 2014;43(2):93-104. doi: 10.1080/16506073.2013.846401. Epub 2013 Nov 12. PMID 24215278